CLINICAL TRIAL: NCT03253679
Title: A Phase 2 Study of AZD1775, a Wee1 Inhibitor, in Patients With CCNE1 Amplification
Brief Title: AZD1775 in Treating Patients With Advanced Refractory Solid Tumors With CCNE1 Amplification
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-01498; NCI-2017-01498 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI10136; 10136 (Other: University of Texas MD Anderson Cancer Center LAO); 10136 (Other: CTEP); UM1CA186688 (NIH)
Record Dates: First submitted 2017-08-17; First posted 2017-08-18 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-09

CONDITIONS: Advanced Malignant Solid Neoplasm; Refractory Malignant Solid Neoplasm
MeSH Terms: interventions — adavosertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (adavosertib) (Experimental): Patients receive adavosertib PO QD on days 1-5 and 8-12. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Adavosertib

INTERVENTIONS:
Drug: Adavosertib — Given PO
  Other Names: AZD-1775; AZD1775; MK-1775; MK1775

SUMMARY:
This phase II trial studies how well AZD1775 works in treating patients with solid tumors with CCNE1 amplification that have spread to other places in the body (advanced) and do not respond to treatment (refractory). AZD1775 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the proportion of patients with the objective response rate (ORR) to adavosertib (AZD1775) in patients with advanced refractory cancers with CCNE1 amplification.

SECONDARY OBJECTIVES:

I. To evaluate the proportion of patients alive and progression free at 6 months of treatment with AZD1775 in patients with advanced refractory cancers with CCNE1 amplification.

II. To evaluate proportion of patients with extended time to progression (time to progression on AZD1775/ time to progression on last line of therapy >= 1.3).

III. To evaluate time until death or disease progression. IV. To identify potential predictive biomarkers beyond the genomic alteration by which treatment is assigned or resistance mechanisms using additional genomic, ribonucleic acid (RNA), protein and imaging-based assessment platforms.

OUTLINE:

Patients receive adavosertib orally (PO) once daily (QD) on days 1-5 and 8-12. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have one of the histologically advanced solid tumors harboring CCNE1 amplification: Their diseases are refractory to, or do not have, standard-of-care therapy; or they declined standard-of-care therapy; CCNE1 amplification is defined in a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory: CCNE1 amplification > 7 based on targeted custom Ampliseq panel on the Ion Torrent Personal Genoma Machine (PGM); or CCNE1 amplification on alternate CLIA platforms such as Foundation One, University of Washington (UW)-OncoPlex-Cancer Gene Panel, Memorial Sloan Kettering (MSK)-Integrated Mutation Profiling of Actionable Cancer Targets (IMPACT), Solid Tumor Genomic Assay (Life Technologies), etc. will also be eligible to be treated after principal investigator (PI) approval; patients with known CCNE1 amplification on local or commercial platforms can start treatment after planned biopsy or submission of recent archival sample; central next generation sequencing (NGS) CCNE1 and fluorescence in-situ hybridization (FISH) testing will be performed to confirm the result
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Has read and understands the informed consent form (ICF) and has given written ICF prior to any study procedures; patients with impaired decision making capacity (IDMC) must have a close caregiver or legally authorized representative (LAR)
* Any prior radiation must have been completed at least 7 days prior to the start of study drugs, and patients must have recovered from any acute adverse effects prior to the start of study treatment
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1
* Absolute neutrophil count (ANC) >= 1500/uL (within 14 days of study drug[s] initiation)
* Hemoglobin (HgB) >= 9 g/dL for mono-therapy (within 14 days of study drug[s] initiation)
* Platelets >= 100,000/uL (within 14 days of study drug[s] initiation)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x upper limit of normal (ULN) or =< 5 x ULN if known hepatic metastases (within 14 days of study drug[s] initiation)
* Serum bilirubin < ULN or < 1.5 x ULN in patients with liver metastases; or total bilirubin < 3.0 x ULN with direct bilirubin within normal limits (WNL) in patients with well documented Gilbert's syndrome (within 14 days of study drug[s] initiation)
* Serum creatinine =< 1.5 x ULN, or calculated creatinine clearance (CrCl) >= 45 mL/min as calculated by the Cockcroft-Gault method or 24-hour measured urine CrCl >= 45 mL/min (within 14 days of study drug[s] initiation)
* Female patients who are not of child-bearing potential and fertile females of childbearing potential who agree to use adequate contraceptive measures from 2 weeks prior to the study and until 1 month after study treatment discontinuation, who are not breastfeeding, and who have a negative serum or urine pregnancy test within 3 days prior to the start of study treatment; male patients willing to abstain or use barrier contraception (i.e. condoms) for the duration of the study and for 3 months after treatment stops
* Willingness and ability to comply with study and follow-up procedures
* Ability to take oral medications without medical history of malabsorption or other chronic gastrointestinal disease, or other conditions that may hamper compliance and/or absorption of the study agent
* No prior treatment with wee1 kinase inhibition
* Provision of an archival tissue block, or 10 formalin-fixed paraffin-embedded (FFPE) slides, if available, and if not available having biopsiable disease and agreeing to pre-treatment biopsies

Exclusion Criteria:

* Use of anti-cancer treatment drug =< 21 days or 5 half-lives (whichever is shorter) prior to the first dose of AZD1775; for drugs for which 5 half-lives is =< 21 days, a minimum of 10 days between termination of the prior treatment and administration of AZD1775 treatment is required
* Previous radiation therapy completed =< 7 days prior to the start of study drugs
* Major surgical procedures =< 28 days of beginning AZD1775, or minor surgical procedures =< 7 days; no waiting period required following port-a-cath or other central venous access placement
* Unresolved grade 2 toxicity from prior therapy (except alopecia or anorexia)
* Patient has an inability to swallow oral medications; Note: Patient may not have a percutaneous endoscopic gastrostomy (PEG) tube or be receiving total parenteral nutrition (TPN)
* No other anticancer-therapy (chemotherapy, immunotherapy, hormonal anti-cancer therapy, radiotherapy [except for palliative local radiotherapy]), biological therapy or other novel agent is to be permitted while the patient is receiving study medication; patients on luteinizing hormone-releasing hormone (LHRH) analogue treatment for more than 6 months are allowed entry into the study and may continue at the discretion of the investigator
* Known malignant central nervous system (CNS) disease other than neurologically stable, treated brain metastases - defined as metastasis having no evidence of progression or hemorrhage for at least 2 weeks after treatment; must be off any systemic corticosteroids for the treatment of brain metastases for at least 14 days prior to enrolment
* Patient has had prescription or non-prescription drugs or other products known to be sensitive to CYP3A4 substrates or CYP3A4 substrates with a narrow therapeutic index, or to be moderate to strong inhibitors/inducers of CYP3A4 which cannot be discontinued 2 weeks prior to day 1 of dosing and withheld throughout the study until 2 weeks after the last dose of study drug; co-administration of aprepitant or fosaprepitant during this study is prohibited; the use of sensitive substrates of CYP3A4, such as atorvastatin, simvastatin and lovastatin, is also prohibited in this study
* Herbal preparations are not allowed throughout the study; these herbal medications include but are not limited to: St. John's wort, kava, ephedra (ma hung), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto and ginseng; patients should stop using these herbal medications 7 days prior to first dose of study treatment
* Any known hypersensitivity or contraindication to the components of the study drug AZD1775
* Any of the following cardiac diseases currently or within the last 6 months as defined by New York Heart Association (NYHA) >= class 2

  * Unstable angina pectoris
  * Congestive heart failure
  * Acute myocardial infarction
  * Conduction abnormality not controlled with pacemaker or medication
  * Significant ventricular or supraventricular arrhythmias (patients with chronic rate-controlled atrial fibrillation in the absence of other cardiac abnormalities are eligible)
* Mean resting corrected QTc interval using the Fridericia formula (QTcF) > 450 msec/male and > 470 msec/female (as calculated per institutional standards) obtained from 3 electrocardiograms (ECGs) 2-5 minutes apart at study entry, or congenital long QT syndrome
* Pregnant or breastfeeding women
* Serious active infection at the time of study entry, or another serious underlying medical condition that would impair the ability of the patient to receive study treatment
* Symptomatic and uncontrolled metastasis in the central nervous system or leptomeningeal or lymphangitic carcinomatosis
* Presence of other active invasive cancers that do not harbor CCNE1 amplification
* Grade 2 or higher peripheral neuropathy
* Human immunodeficiency virus requiring highly active antiretroviral therapy (HAART) treatment due to unknown drug-drug interactions or has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive or C virus [e.g., hepatitis C virus (HCV) RNA (quantitative) is detected]) infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Siqing Fu, Principal Investigator — University of Texas MD Anderson Cancer Center LAO
Locations (9):
- United States (9):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of Colorado Hospital, Aurora, Colorado
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Fu S, Yao S, Yuan Y, Previs RA, Elias AD, Carvajal RD, George TJ, Yuan Y, Yu L, Westin SN, Xing Y, Dumbrava EE, Karp DD, Piha-Paul SA, Tsimberidou AM, Ahnert JR, Takebe N, Lu K, Keyomarsi K, Meric-Bernstam F. Multicenter Phase II Trial of the WEE1 Inhibitor Adavosertib in Refractory Solid Tumors Harboring CCNE1 Amplification. J Clin Oncol. 2023 Mar 20;41(9):1725-1734. doi: 10.1200/JCO.22.00830. Epub 2022 Dec 5. PMID 36469840

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Adavosertib): Participants receive adavosertib PO QD on days 1-5 and 8-12. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Adavosertib)
Started | 31
Completed | 30
Not Completed | 1
Not completed — Screen Failure | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Adavosertib)
Number analyzed (Participants) | 30
Age, Continuous [Mean (Inter-Quartile Range); unit: Years] — Population: One participant did not receive any study agent. Thus, 30 patients were considered evaluable
  Years | 65 [42 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: One participant did not receive any study agent. Thus, 30 patients were considered evaluable.
  Participants
    Hispanic or Latino | 4
    Not Hispanic or Latino | 26
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: One participant did not receive any study agent. Thus, 30 patients were considered evaluable
  Participants
    American Indian or Alaska Native | 0
    Asian | 3
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 2
    White | 25
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as a complete response or partial response and consistent with Response Evaluation Criteria in Solid Tumors version 1.1 criteria. The ORR rate will be compared against a null benchmark value of 5%.
Time Frame: Up to 2 years 6 months
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Treatment (Adavosertib)
Number analyzed (Participants) | 30
percentage | 27 [12 to 46]

2. Secondary Outcome: To Evaluate the Proportion of Patients Alive and Progression Free of Treatment With AZD1775 in Patients With Advanced Refractory Cancers With CCNE1 Amplification.
Description: Estimated using the Kaplan-Meier Method.
Time Frame: Up to 2 years 6 months
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Treatment (Adavosertib)
Number analyzed (Participants) | 30
percentage | 37 [20 to 56]

3. Secondary Outcome: To Evaluate Time Until Death or Disease Progression.
Description: Estimated using the Kaplan-Meier Method.
Time Frame: Up to 2 years 6 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Adavosertib)
Number analyzed (Participants) | 30
Months | 9.9 [4.8 to 15]

4. Secondary Outcome: Duration of Responses
Description: (time to progression on AZD1775/ time to progression on last line of therapy >= 1.3).
Time Frame: Up to 2 years 6 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Adavosertib)
Number analyzed (Participants) | 30
Months | 4.1 [1.8 to 6.4]

5. Secondary Outcome: Identify Potential Predictive Biomarkers Beyond the Genomic Alteration by Which Treatment is Assigned or Resistance Mechanisms Using Additional Genomic, RNA, Protein and Imaging-based Assessment Platforms.
Description: Immunohistochemistry, reverse phase protein arrays, and next generation sequencing for targeted exome panel are used to reveal potential biomarkers predicting major clinical outcomes, and potential mechanisms of acquired resistance by comparing molecular signatures at baseline versus at time of relapse in responders.
Time Frame: Up to 2 years 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Adavosertib)
Number analyzed (Participants) | 30
Participants
  TP53 gene aberration | 27
  AKT2 amplification | 7
  MYC amplification | 5
  CCND2 amplification | 3
  NOTCH1 mutation | 3

ADVERSE EVENTS:
Time Frame: Up to 2 years 6 months
Arm/Group | Treatment (Adavosertib)
All-Cause Mortality (participants affected / at risk) | 3/30
Serious Adverse Events (participants affected / at risk) | 20/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Adavosertib) (N=30)
Dehydration (Metabolism and nutrition disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Fatigue (General disorders) | 2
Thromboemolic event (Vascular disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Fever (General disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 — small bowel obstruction
Nausea (Gastrointestinal disorders) | 1
Acute kidney failure (Renal and urinary disorders) | 1
Sepsis (Infections and infestations) | 1
Delirium (Nervous system disorders) | 1
Portal vein thrombosis (Vascular disorders) | 1
Depression (Nervous system disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Non-hemolytic transfusion reaction (General disorders) | 1
Bladder infection (Infections and infestations) | 1
Renal failure (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Skin infection (Infections and infestations) | 1
Blood bilirubin increased (Investigations) | 1
Confusion (Nervous system disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Creatinine increased (Investigations) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Disease progression (General disorders) | 1
Enterocolitis infections (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Adavosertib) (N=30)
Abdominal pain (Gastrointestinal disorders) | 16
ALP increased (Investigations) | 9
ALT increased (Investigations) | 7
Anemia (Blood and lymphatic system disorders) | 26
Anorexia (Metabolism and nutrition disorders) | 9
AST increased (Investigations) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 11
Constipation (Gastrointestinal disorders) | 12
Creatinine increased (Investigations) | 5
Dehydration (Metabolism and nutrition disorders) | 4
Diarrhea (Gastrointestinal disorders) | 28
Dizziness (Nervous system disorders) | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9
Edema limbs (General disorders) | 15
Fatigue (General disorders) | 20
Headache (Nervous system disorders) | 7
Hyperglycemia (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 20
Hypocalcemia (Metabolism and nutrition disorders) | 10
Hyponatremia (Metabolism and nutrition disorders) | 14
Lymphocyte count decreased (Investigations) | 12
Nausea (Gastrointestinal disorders) | 25
Neutrophil count decreased (Investigations) | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Platelet count decreased (Investigations) | 25
Vomiting (Gastrointestinal disorders) | 12
WBC decreased (Investigations) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-02): https://cdn.clinicaltrials.gov/large-docs/79/NCT03253679/Prot_SAP_000.pdf